CLINICAL TRIAL: NCT00963040
Title: The Effect of Intranasal Oxytocin on Headache Intensity and Headache-associated Symptoms in Patients Suffering From Chronic Daily Headache
Brief Title: Effect of Intranasal Oxytocin on Headache in Chronic Daily Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedVadis Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TI-004, TI-005
Record Dates: First submitted 2009-08-18; First posted 2009-08-20 (Estimated); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Chronic Daily Headache
Keywords: intranasal oxytocin; acute headache treatment; chronic daily headache
MeSH Terms: conditions — Headache Disorders | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Syntocinon® TI-004 protocol (Experimental): Treated group
  Interventions: Drug: Syntocinon
- Sterile water TI-004 protocol (Placebo Comparator): Placebo group
  Interventions: Drug: Sterile water
- Syntocinon® TI-005 protocol (Experimental)
  Interventions: Drug: Syntocinon
- Sterile water TI-005 protocol (Placebo Comparator)
  Interventions: Drug: Sterile water

INTERVENTIONS:
Drug: Syntocinon — 4 actuations in each nostril for a total dose of 32 IU
  Other Names: Oxytocin
  Arms: Syntocinon® TI-004 protocol
Drug: Sterile water — 4 actuations in each nostril
  Other Names: Placebo
  Arms: Sterile water TI-004 protocol
Drug: Syntocinon — 8 actuations in each nostril for a total dose of 64 IU
  Other Names: Oxytocin
  Arms: Syntocinon® TI-005 protocol
Drug: Sterile water — 8 actuations in each nostril
  Other Names: Placebo
  Arms: Sterile water TI-005 protocol

SUMMARY:
The objective of this prospective, randomized, double-blind, parallel-group, placebo-controlled study is to determine the effectiveness of intranasal oxytocin in subjects suffering from chronic daily headache.

DETAILED DESCRIPTION:
The TI004 and TI005 studies both used a randomized, double-blind, placebo-controlled, parallel-group study design. A protocol-specified interim analysis was performed after completion of the first 40 subjects, resulting in termination of the TI004 study and development of the TI005 protocol, which included the following changes from the TI004 protocol:

1. Increase in oxytocin dose from 32 to 64 IU;
2. Extension of the in-clinic observation period from 2 hours post-dose to 4-hours post-dose;
3. Reduction in sample size from 40 to 20 subjects;
4. Elimination of the laboratory measurements during the screening visit, allowing V1 and V2 potentially to be combined, expediting study completion;
5. Adding in-clinic observation and assessment at 3 hours and 4 hours post-dose and out-of-clinic assessment at 8 hours post-dose.

The primary outcome measure is the reduction in headache intensity after drug administration; secondary outcome measures are the headache symptoms, nausea, vomiting, photophobia, and phonophobia. Additional secondary outcome measures are intake of rescue medication and patient satisfaction over a period of 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Headache on equal to or more than 15 days per month for at least 6 months; the headaches can be migraine or tension.
2. More than half of the monthly headaches are of moderate or severe intensity on the 4-point categorical pain rating scale and are assessed as 6 or higher on the 11-point numerical pain rating scale.
3. Headaches typically last for at least 4 hours.
4. Subjects are on a stable headache treatment, if any, for at least 2 months.

Exclusion Criteria:

1. Headache symptoms assessed to be predominately occipital.
2. Allergy to oxytocin.
3. History of addictive behavior (e.g. alcoholism, drug abuse).
4. History of significant psychiatric disorder.
5. History of clinically-significant, functionally-impairing cardiovascular or pulmonary disease.
6. Upper-respiratory tract infection at the time of randomization.
7. Past or current history of any condition that may hinder study procedures or confuse interpretation of data.
8. Nasal obstruction of any cause as determined at screening.
9. Major surgery or trauma within 4 weeks of screening.
10. Women who are pregnant as evidenced by a serum HCG, nursing, or trying to conceive.
11. Use of intranasally administered medications, for example, vasoconstrictors or corticosteroids, within 2 weeks of randomization.
12. Use of an investigational medication or device within 30 days of randomization.
13. Unable or unwilling to adhere to the study-specific procedures and restrictions.
14. Any condition that in the opinion of the investigator would compromise the safety of the subject or the quality of the data.
15. Alanine aminotransaminase (ALT) or aspartate aminotransaminase (AST) equal or greater than 3 times the upper limit of normal (ULN).
16. Serum creatinine of equal or greater than 1.8 mg/dL. Resting, sitting systolic blood pressure equal or greater than 160 mmHg or diastolic blood pressure equal or greater than 100 mmHg at screening. For patients with previously diagnosed hypertension, antihypertensive medications must be stable for at least 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Egilius LH Spierings, MD, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- MedVadis Research Corporation, Wellesley Hills, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited at dedicated research center
Pre-assignment Details: In total 79 subjects were screened, of which five were screen failures in the strict sense of the word and 14 were not randomized because the 6-week treatment period had elapsed.
Groups:
- Syntocinon® (Oxytocin) TI-004 Protocol: Self-administered by participants in the upright sitting position with the neck flexed. The pump was primed and one nostril was closed with the finger. The tip of the bottle was inserted into the other nostril at an angle of 60 degrees. One actuation (4 IU) was administered while gently sniffing through that nostril. The tip of the bottle was then inserted into the other nostril for administration of another 4 IU. This procedure was repeated three times with 5-minute intervals (allowing for medication uptake and clearance) for a total dose of 32 IU followed by in-clinic observation for 2 hours post-dose in the TI004 study
- Placebo TI-004 Protocol: Administration of placebo similar to oxytocin arm: 4 actuations in each nostril of sterile water with in-clinic observation for 2 hours post-dose in the TI004 study
- Syntocinon® (Oxytocin) TI-005 Protocol: Self-administered by participants in the upright sitting position with the neck flexed. The pump was primed and one nostril was closed with the finger. The tip of the bottle was inserted into the other nostril at an angle of 60 degrees. One actuation (4 IU) was administered while gently sniffing through that nostril. The tip of the bottle was then inserted into the other nostril for administration of another 4 IU. This procedure was repeated seven times with 5-minute intervals (allowing for medication uptake and clearance) for a total dose of 64 IU followed by 4 hours post-dose in-clinic observation in the TI005 study.
- Placebo TI-005 Protocol: Administration of placebo similar to oxytocin arm: 7 actuations of sterile with 5-minute intervals followed by 4 hours post-dose of in-clinic observation in the TI005 study.
Period: TI-004 Protocol
Arm/Group | Syntocinon® (Oxytocin) TI-004 Protocol | Placebo TI-004 Protocol | Syntocinon® (Oxytocin) TI-005 Protocol | Placebo TI-005 Protocol
Started | 22 | 18 | 0 | 0
Completed | 22 | 18 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: TI-005 Protocol
Arm/Group | Syntocinon® (Oxytocin) TI-004 Protocol | Placebo TI-004 Protocol | Syntocinon® (Oxytocin) TI-005 Protocol | Placebo TI-005 Protocol
Started | 0 | 0 | 12 | 8
Completed | 0 | 0 | 12 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Syntocinon® (Oxytocin) TI-004 Protocol: 32 IU intranasally
- Placebo TI-004 Protocol; Placebo TI-005 Protocol: Sterile water intranasally
- Syntocinon® (Oxytocin) TI-005 Protocol: 64 IU intranasally
- Total: Total of all reporting groups
Arm/Group | Syntocinon® (Oxytocin) TI-004 Protocol | Placebo TI-004 Protocol | Syntocinon® (Oxytocin) TI-005 Protocol | Placebo TI-005 Protocol | Total
Number analyzed (Participants) | 22 | 18 | 12 | 8 | 60
Age, Continuous [Mean (Standard Deviation); unit: years]
  Protocol TI-004 | 44.5 (11.37) | 41.0 (9.4) | NA (NA) — Data for TI-004 only | NA (NA) — Data for TI-004 only | 42.9 (10.6)
  Protocol TI-005 | NA (NA) — Data for TI-005 only | NA (NA) — Data for TI-005 only | 45.0 (10.8) | 39.5 (15.1) | 42.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 6 | 3 | 36
  Male | 7 | 6 | 6 | 5 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 0 | 3
  Not Hispanic or Latino | 20 | 17 | 12 | 8 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 5 | 0 | 0 | 13
  White | 12 | 10 | 0 | 0 | 22
  More than one race | 2 | 3 | 0 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Headache Intensity
Description: Number (Percentage) of participants with headache improvement defined as a reduction from moderate or severe to mild or absent (4-point categorical scale)
Time Frame: 2 hours after administration of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Syntocinon® (Oxytocin) TI-004 Protocol | Placebo TI-004 Protocol | Syntocinon® (Oxytocin) TI-005 Protocol | Placebo TI-005 Protocol
Number analyzed (Participants) | 22 | 18 | 12 | 8
Participants | 6 | 4 | 1 | 3

2. Secondary Outcome: Reduction in Headache Intensity
Description: as for outcome 1
Time Frame: ½, 1, 3 (TI005 study only), 4, 8 (TI005 study only), and 24 hours after administration of study medication
Population: Number of participants analyzed indicates the number of participants available at each time point. 3 hours and 8 hours were not collected for TI-004 protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Syntocinon® (Oxytocin) TI-004 Protocol | Placebo TI-004 Protocol | Syntocinon® (Oxytocin) TI-005 Protocol | Placebo TI-005 Protocol
Number analyzed (Participants) | 22 | 18 | 12 | 8
Participants
  0.5 hours after administration | 0 | 1 | 0 | 0
  1 hour after administration | 3 | 1 | 0 | 1
  3 hours after administration: number analyzed (Participants) | 0 | 0 | 12 | 8
  3 hours after administration |  |  | 1 | 4
  4 hours after administration: number analyzed (Participants) | 22 | 17 | 12 | 8
  4 hours after administration | 11 | 2 | 4 | 5
  8 hours after administration: number analyzed (Participants) | 0 | 0 | 12 | 8
  8 hours after administration |  |  | 4 | 5
  24 hours after administration | 10 | 7 | 6 | 6

3. Secondary Outcome: Average Headache Intensity
Description: Average headache intensity as rated on the 11-point numerical rating scale (0 = no pain; 10 = worst pain possible).
Time Frame: ½, 1, 2, 3 (TI005 study only), 4, 8 (TI005 study only), and 24 hours after administration of study medication
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Syntocinon® (Oxytocin) TI-004 Protocol | Placebo TI-004 Protocol | Syntocinon® (Oxytocin) TI-005 Protocol | Placebo TI-005 Protocol
Number analyzed (Participants) | 22 | 18 | 12 | 8
score on a scale
  0.5 hours after administration | 7.1 (1.5) | 7.1 (1.6) | 6.5 (0.8) | 6.1 (1.2)
  1 hour after administration | 6.2 (2.3) | 6.5 (1.3) | 6.1 (1.1) | 5.7 (1.8)
  2 hours after administration | 5.8 (2.2) | 5.9 (1.7) | 5.7 (1.1) | 4.6 (1.9)
  3 hours after administration: number analyzed (Participants) | 0 | 0 | 12 | 8
  3 hours after administration |  |  | 4.8 (1.7) | 3.5 (2.1)
  4 hours after administration | 3.8 (2.9) | 6.0 (1.9) | 3.9 (2.6) | 2.8 (2.2)
  8 hours after administration: number analyzed (Participants) | 0 | 0 | 12 | 8
  8 hours after administration |  |  | 4.3 (2.5) | 3.0 (2.3)
  24 hours after administration | 4.2 (2.8) | 4.5 (3.0) | 3.5 (3.0) | 1.8 (2.8)

4. Secondary Outcome: Presence of Nausea, Vomiting, Photophobia, and Phonophobia
Description: Number (percentage) of participants with effects of oxytocin on symptoms associated with chronic daily headache, such as nausea, vomiting, photophobia, and phonophobia
Time Frame: ½, 1, 2, 3 (TI005 study only), 4, 8 (TI005 study only), and 24 hours after administration of study medication
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Syntocinon® (Oxytocin) TI-004 Protocol | Placebo TI-004 Protocol | Syntocinon® (Oxytocin) TI-005 Protocol | Placebo TI-005 Protocol
Number analyzed (Participants) | 22 | 18 | 12 | 8
Participants
  Nausea at 0.5 hours | 7 | 2 | 0 | 1
  Nausea at 1 hour | 5 | 3 | 0 | 1
  Nausea at 2 hours | 3 | 2 | 1 | 2
  Nausea at 3 hours: number analyzed (Participants) | 0 | 0 | 12 | 8
  Nausea at 3 hours |  |  | 0 | 1
  Nausea at 4 hours | 2 | 6 | 0 | 0
  Nausea at 8 hours: number analyzed (Participants) | 0 | 0 | 12 | 8
  Nausea at 8 hours |  |  | 1 | 1
  Nausea at 24 hours | 2 | 2 | 0 | 0
  Vomiting at 0.5 hours | 1 | 0 | 0 | 0
  Vomiting at 1 hour | 0 | 0 | 0 | 0
  Vomiting at 2 hours | 1 | 0 | 0 | 0
  Vomiting at 3 hours: number analyzed (Participants) | 0 | 0 | 12 | 8
  Vomiting at 3 hours |  |  | 0 | 0
  Vomiting at 4 hours | 0 | 2 | 0 | 0
  Vomiting at 8 hours: number analyzed (Participants) | 0 | 0 | 12 | 8
  Vomiting at 8 hours |  |  | 0 | 0
  Vomiting at 24 hours | 0 | 0 | 0 | 0
  Photophobia at 0.5 hours | 17 | 15 | 6 | 3
  Photophobia at 1 hour | 14 | 13 | 4 | 2
  Photophobia at 2 hours | 10 | 13 | 4 | 1
  Photophobia at 3 hours: number analyzed (Participants) | 0 | 0 | 12 | 8
  Photophobia at 3 hours |  |  | 5 | 1
  Photophobia at 4 hours | 7 | 14 | 4 | 1
  Photophobia at 8 hours: number analyzed (Participants) | 0 | 0 | 12 | 8
  Photophobia at 8 hours |  |  | 3 | 1
  Photophobia at 24 hours | 9 | 7 | 4 | 0
  Phonophobia at 0.5 hours | 11 | 10 | 6 | 2
  Phonophobia at 1 hour | 10 | 12 | 3 | 1
  Phonophobia at 2 hours | 10 | 9 | 3 | 1
  Phonophobia at 3 hours: number analyzed (Participants) | 0 | 0 | 12 | 8
  Phonophobia at 3 hours |  |  | 3 | 1
  Phonophobia at 4 hours | 6 | 10 | 2 | 1
  Phonophobia at 8 hours: number analyzed (Participants) | 0 | 0 | 12 | 8
  Phonophobia at 8 hours |  |  | 2 | 1
  Phonophobia at 24 hours | 4 | 5 | 3 | 0

5. Secondary Outcome: Intake of Rescue Medication
Description: Number of participants who took rescue medication (examples: ibuprofen, Tylenol, zolmitriptan) for headache at any time within the 24 hours after intervention administration.
Time Frame: Up to 24 hours after intervention administration
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Syntocinon® (Oxytocin) TI-004 Protocol | Placebo TI-004 Protocol | Syntocinon® (Oxytocin) TI-005 Protocol | Placebo TI-005 Protocol
Number analyzed (Participants) | 22 | 18 | 12 | 8
Participants | 12 | 10 | 4 | 2

6. Secondary Outcome: Participant Satisfaction
Description: Participants rated their satisfaction with treatment on a 4-point scale as "Excellent", "Good", "Moderate", or "Poor". Number (percentage) of participants who reported each rating.
Time Frame: Up to 24 hours after intervention administration
Measure: Count of Participants; unit: Participants
Arm/Group | Syntocinon® (Oxytocin) TI-004 Protocol | Placebo TI-004 Protocol | Syntocinon® (Oxytocin) TI-005 Protocol | Placebo TI-005 Protocol
Number analyzed (Participants) | 22 | 18 | 12 | 8
Participants
  "Excellent" satisfaction rating | 4 | 5 | 4 | 2
  "Good" satisfaction rating | 7 | 5 | 4 | 5
  "Moderate" satisfaction rating | 6 | 4 | 2 | 0
  "Poor" satisfaction rating | 4 | 2 | 2 | 1
  Satisfaction rating not reported | 1 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Safety was monitored through the collection of health-status changes and adverse-event occurrences during the 8-week study
Description: AEs were recorded with date of onset and resolution, intensity, and relationship to study medication. The safety analysis was conducted on the intention-to-treat population, including all subjects assigned through randomization to treatment with oxytocin or placebo.
Groups:
- Sterile Water TI-004 Protocol: Administration of placebo similar to oxytocin arm: 4 actuations in each nostril of sterile water with in-clinic observation for 2 hours post-dose in the TI004 study
- Sterile Water TI-005 Protocol: Administration of placebo similar to oxytocin arm: 7 actuations of sterile with 5-minute intervals followed by 4 hours post-dose of in-clinic observation in the TI005 study.
Arm/Group | Syntocinon® (Oxytocin) TI-004 Protocol | Sterile Water TI-004 Protocol | Syntocinon® (Oxytocin) TI-005 Protocol | Sterile Water TI-005 Protocol
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18 | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18 | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 8/22 | 3/18 | 2/12 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Syntocinon® (Oxytocin) TI-004 Protocol (N=22) | Sterile Water TI-004 Protocol (N=18) | Syntocinon® (Oxytocin) TI-005 Protocol (N=12) | Sterile Water TI-005 Protocol (N=8)
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 — Treatment-related adverse event: Assessed by the investigator as possibly or probably causally related to treatment
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 0 — Treatment-related adverse event: Assessed by the investigator as possibly or probably causally related to treatment
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 — NOT Treatment-related adverse event: Assessed by the investigator as not related to treatment
Rhinitis (Infections and infestations) | 2 | 0 | 0 | 0 — Treatment-related adverse event: Assessed by the investigator as possibly or probably causally related to treatment
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 — NOT Treatment-related adverse event: Assessed by the investigator as not related to treatment
Ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 — NOT Treatment-related adverse event: Assessed by the investigator as not related to treatment
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 — Treatment-related adverse event: Assessed by the investigator as possibly or probably causally related to treatment
Agitation (Nervous system disorders) | 1 | 0 | 0 | 0 — Treatment-related adverse event: Assessed by the investigator as possibly or probably causally related to treatment
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Treatment-related adverse event: Assessed by the investigator as possibly or probably causally related to treatment
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Treatment-related adverse event: Assessed by the investigator as possibly or probably causally related to treatment
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Treatment-related adverse event: Assessed by the investigator as possibly or probably causally related to treatment
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 — NOT Treatment-related adverse event: Assessed by the investigator as not related to treatment
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 — NOT Treatment-related adverse event: Assessed by the investigator as not related to treatment
Light headedness (Nervous system disorders) | 0 | 1 | 0 | 0 — Treatment-related adverse event: Assessed by the investigator as possibly or probably causally related to treatment
Ankle sprain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 — NOT Treatment-related adverse event: Assessed by the investigator as not related to treatment
Nasal irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Treatment-related adverse event: Assessed by the investigator as possibly or probably causally related to treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No